CLINICAL TRIAL: NCT01018407
Title: Multisite Randomized Control Treatment of Early Intervention for Spoken Communication in Autism
Brief Title: Interventions for Communication in Autism Network
Acronym: ICAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Connie Kasari, Ph.D., Professor of Psychological Studies in Education and Psychiatry, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01MH084864-01A109; 1R01MH084864 (NIH); DDTR B2-MBA (Other Grant/Funding Number: National Institute of Mental Health)
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Discrete Trial Training (Experimental): Targets nonverbal imitation, match-to-sample, verbal imitation, imitation of play activities, receptive language, and expressive language. 5 hours per week of individual instruction for 4 months (Two 30-minute sessions per day, five days per week) with reductions in classroom pull out sessions in months 5 and 6 with implementation of 1 hour per week of in-home parent training for the last 2 months.
  Interventions: Behavioral: Discrete Trial Training
- Interpersonal Developmental Approach (Experimental): Targets Joint Attention and Symbolic Play. 5 hours per week of individual instruction for 4 months (Two 30-minute sessions per day, five days per week) with reductions in classroom pull out sessions in months 5 and 6 with implementation of 1 hour per week of in-home parent training for the last 2 months.
  Interventions: Behavioral: Interpersonal Developmental Approach

INTERVENTIONS:
Behavioral: Discrete Trial Training — UCLA model, developed by Lovaas and colleagues (Smith, Groen & Wynn, 2000). Two 30-minute sessions daily (5 hours/week) of 1:1 intervention focusing on imitation, match-to-sample, receptive and expressive language. Using operant conditioning, the therapist works individually with a child in a distraction-free setting and administers approximately 10 trials in a sitting, with breaks between sittings.
  During months 5 and 6, we will provide parents with training in an apprenticeship format one day per week for an hour per day. The clinician will demonstrate a DTT instructional program, then the parent will take a turn implementing it. The clinician and parent will give each other feedback on their implementation of the program.
  Other Names: DTT
  Arms: Discrete Trial Training
Behavioral: Interpersonal Developmental Approach — Focus on teaching joint attention and symbolic play developmentally via floor play milieu teaching approach. Principles applied include following the child's lead and interest in activities, talking about what the child is doing, repeating back what the child says, expanding on what child says, giving corrective feedback, sitting close to the child and making eye-contact, and making environmental adjustments to engage the child (Kasari et al., 2006).
  Parents will be incorporated into the treatment to encourage joint engagement with their child and to focus specifically on joint attention and play skills in their interactions. Each home session will last one hour (once a week) during month 5 and 6 and will involve therapist modeling, and coaching of parent in child-directed activities.
  Other Names: IDA
  Arms: Interpersonal Developmental Approach

SUMMARY:
The goal of this project is to compare the efficacy of two interventions for improving spoken language and reducing symptoms of autism.

DETAILED DESCRIPTION:
While significant progress has been made toward identifying effective interventions for preschool-age children with autism (National Research Council, 2001), few scientifically rigorous studies have compared active ingredients of these interventions or examined outcomes focused on core deficits. To address these areas of need, this collaborative, multi-site project combines the expertise of investigators experienced in randomized controlled clinical trials (RCTs), in the study of core deficits in young children with autism, and in data management and analysis of multi-site clinical trials.

The goal of this project is to compare the efficacy of two interventions for improving spoken language and reducing symptoms of autism: (1) Discrete trial training (DTT)--an applied behavior analysis approach emphasizing highly structured teaching of school readiness skills (match-to-sample, imitation, functional play, and receptive and expressive language) and (2) Interpersonal developmental approach (IDA): a visually supported, child-focused, flexible engagement, social communicative engagement approach on joint attention, symbolic play, and the use of conventional symbols within socially valid communicative contexts.

Children will be randomly assigned to DTT or IDA. In each condition, children's ongoing early intervention programs will be augmented with two 30-minute sessions daily of the study intervention (DTT or IDA) conducted by supervised therapists for 4 months, with transition to home therapy for 2 months.

Potential moderators (e.g., initial mental age and language age) and mediators (e.g. parent synchronization of joint attention and changes in parental expectancies) on treatment outcome will also be examined.

The assessment measures will include diagnostic and developmental measures. There are three sets of assessments. The first set of assessments is to determine whether the child is eligible for the study. If the child is eligible, we will complete the next set of assessments, which are completed at three points: (1) prior to entry into the treatment (this is a baseline measurement conducted just before the start of the treatment phase); (2) at exit; and (3) at a 6 month follow-up. Several assessments will also be completed after 2 months, 4 months, and 6 months.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of an autism spectrum disorder (Autistic Disorder or Pervasive Developmental Disorder Not Otherwise Specified) from a licensed doctoral-level clinician, confirmed by the Autism Diagnostic Observation Schedule and clinical judgment.
2. Chronological age between 33 and 54 months
3. Must be receiving at least 12.5 hours per week of early intervention or preschool developmental services, some of which must be provided in a school setting.
4. Cognitive and language requirements (at least two of the following three criteria must be met:

   * >12 months for visual reception (as determined by Mullen Scales of Early Learning) or receptive language (as determined by Mullen or Reynell Developmental Language Scales)
   * a score of 1,2 or 3 on the ADOS Module 1
   * <30 spontaneous communicative words, as determined by behavior assessments (Mother- Child Interaction, Early Social Communication Scales, and Structured Play Assessment)

Exclusion criteria:

1. Major medical conditions other than autism, specifically (a) genetic disorders such as Fragile X, Down syndrome, or tuberous sclerosis, (b) sensory disabilities such as blindness or deafness, and (c) motor disabilities such as cerebral palsy
2. Nonverbal mental age < 12 months, based on a nonverbal score from the Mullen Scales of Early Learning (Mullen, 1995), as reliability of a diagnosis of autism is questionable at this developmental level.
3. Expressive language level that exceeds the First Words level, as evidenced by an age equivalent of 24 months or greater on the Expressive Language Scale of the Reynell
4. Exposure to English less than 50% of the time

Ages: 33 Months to 54 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2009-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Reynell Developmental Language Scale | Pre-treatment, post-treatment, and 6 months later

SECONDARY OUTCOMES:
McArthur-Bates Communicative Development Inventory (Word and Gestures Inventory and/or Words and Sentences Inventory) | Pre-treatment, post-treatment, and 6-month follow up
Caregiver-child Interaction | Pre-treatment, three times during active intervention, post-treatment, and 6-month follow up
Early Social Communication Scale | Pre-treatment, post-treatment, and 6-month follow up
Structured Play Assessment | Pre-treatment, post-treatment, and 6-month follow up

CONTACTS AND LOCATIONS:
Overall Officials: Connie Kasari, PhD, Principal Investigator — University of California, Los Angeles
Locations (3):
- United States (3):
  - University of California, Los Angeles, Los Angeles, California
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Rochester, Rochester, New York

REFERENCES:
- [Background] Kasari C, Freeman S, Paparella T. Joint attention and symbolic play in young children with autism: a randomized controlled intervention study. J Child Psychol Psychiatry. 2006 Jun;47(6):611-20. doi: 10.1111/j.1469-7610.2005.01567.x. PMID 16712638
- [Background] Smith T, Groen AD, Wynn JW. Randomized trial of intensive early intervention for children with pervasive developmental disorder. Am J Ment Retard. 2000 Jul;105(4):269-85. doi: 10.1352/0895-8017(2000)1052.0.CO;2. PMID 10934569
- [Result] Kasari C, Shire S, Shih W, Landa R, Levato L, Smith T. Spoken language outcomes in limited language preschoolers with autism and global developmental delay: RCT of early intervention approaches. Autism Res. 2023 Jun;16(6):1236-1246. doi: 10.1002/aur.2932. Epub 2023 Apr 18. PMID 37070270
- [Result] Brady NC, Romine RES, Holbrook A, Fleming KK, Kasari C. Measuring Change in the Communication Skills of Children With Austim Spectrum Disorder Using the Communication Complexity Scale. Am J Intellect Dev Disabil. 2020 Nov 1;125(6):481-492. doi: 10.1352/1944-7558-125.6.481. PMID 33211817
- [Result] Brady NC, Fleming K, Romine RS, Holbrook A, Muller K, Kasari C. Concurrent Validity and Reliability for the Communication Complexity Scale. Am J Speech Lang Pathol. 2018 Feb 6;27(1):237-246. doi: 10.1044/2017_AJSLP-17-0106. PMID 29383380
- [Result] Pizzano M, Shire S, Shih W, Levato L, Landa R, Lord C, Smith T, Kasari C. Profiles of minimally verbal autistic children: Illuminating the neglected end of the spectrum. Autism Res. 2024 Jun;17(6):1218-1229. doi: 10.1002/aur.3151. Epub 2024 May 27. PMID 38803132
- See also: Related Info — http://www.autism.ucla.edu